CLINICAL TRIAL: NCT00002802
Title: PHASE III MULTICENTRE TRIAL OF TREATMENT OF NEUROBLASTOMA IN CHILDREN AND ADOLESCENTS
Brief Title: Therapy Based on Stage of Disease and Risk Assessment in Treating Children With Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000064902; GER-NB90; EU-96004
Record Dates: First submitted 1999-11-01; First posted 2004-05-12 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Dacarbazine; Doxorubicin; Etoposide; Ifosfamide; Melphalan; Mesna; Vincristine; Vindesine

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: melphalan
Drug: mesna
Drug: vincristine sulfate
Drug: vindesine
Procedure: autologous bone marrow transplantation
Procedure: conventional surgery
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy
Radiation: radioisotope therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which treatment regimen is most effective in treating patients with different stages of and risk factors for neuroblastoma.

PURPOSE: Phase III trial to study the effectiveness of therapy based on stage of disease and risk assessment in treating children with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Increase the survival rates and duration of survival in children and adolescents with neuroblastoma by using stage- and risk group-appropriate therapy. II. Determine whether using cisplatin/etoposide/vindesine and vincristine/dacarbazine/ifosfamide/doxorubicin instead of cisplatin/teniposide and vincristine/dacarbazine/cyclophosphamide/doxorubicin improves remission rate and lessens toxicity in patients with stage 3C, 3D, or 4 neuroblastoma. III. Determine whether local radiotherapy to the primary tumor and bone metastasis improves local tumor control in these patients. IV. Compare the efficacy and survival associated with short-term, high-dose conditioning chemotherapy plus autologous bone marrow transplantation vs. long-term, low-dose cytostatic chemotherapy as consolidation therapy in these patients. V. Determine whether early use of low-dose doxorubicin/vincristine plus hepatic irradiation slows disease progression in patients with stage 4S-C neuroblastoma. VI. Determine whether 4 courses of chemotherapy reduces the occurrence of local and systemic relapse in patients with stages 2, 3A, and 3B neuroblastoma. VII. Determine whether serum tumor markers (LDH, catecholamine metabolites, and neuron-specific enolase) are predictive of remission behavior.

OUTLINE: Patients are staged according to the International Neuroblastoma Staging System and are further defined by progressively less favorable risk groups based on age at diagnosis, serum LDH, and tumor resectability (risk groups A, B, C, and D, representing presence of 0, 1, 2, or 3 risk factors, respectively). Patients who are unable to be resected at entry or with incomplete resection are re-evaluated at 4-month intervals for the appropriateness of tumor resection. STAGE 1 PATIENTS Patients undergo complete primary tumor resection and no other therapy. STAGES 2, 3A, AND 3B PATIENTS Patients undergo primary tumor resection, followed by cisplatin, etoposide, vindesine (PEV) alternating monthly with vincristine, dacarbazine, ifosfamide, doxorubicin (VDIA). Patients in complete remission (CR) discontinue therapy, while those with less than CR receive additional therapy as outlined below for stages 3C, 3D, and 4 patients, except that these patients are not eligible for bone marrow transplantation. STAGES 3C, 3D, AND 4 PATIENTS Patients receive PEV and VDIA as above, with radiotherapy to sites of metastases during the third and fourth courses, following which autologous bone marrow is collected. Following marrow harvest, patients receive up to 4 more alternating courses of PEV/VDIA; those with no response or progressive disease after the sixth chemotherapy course are referred for other therapy. Patients who complete PEV/VDIA receive 3 weeks of radiotherapy to the primary tumor bed or residual tumor. Stage 4 patients in complete or very good partial remission and with sufficient harvested marrow undergo ABMT following radiotherapy. Myeloablation consists of high-dose MIBG radioisotope therapy followed by high-dose melphalan, etoposide, and carboplatin. All other patients and those who refuse ABMT receive 1 year of alternating, low-dose chemotherapy courses, beginning concurrently with initiation of radiotherapy. One regimen consists of oral melphalan/etoposide for 5 days and the other regimen consists of intravenous vincristine on 1 day and oral cyclophosphamide for 7 days. Therapy continues for 1 year. STAGE 4S PATIENTS Patients in risk groups 4S-A and 4S-B receive no therapy. Patients in group 4S-C receive 4-8 weekly injections of doxorubicin and vincristine (AV). Patients with tumor progression may receive low-dose radiotherapy. Primary tumor resection may be delayed up to 8 months after diagnosis in these patients. Use of G-CSF is allowed but not recommended.

PROJECTED ACCRUAL: Approximately 500 patients will be accrued on this multicenter study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Neuroblastoma with diagnosis based on one of the following: Histologic confirmation Cytologic confirmation in bone marrow and elevated catecholamine metabolites Typical tumor appearance on CT, MRI, or ultrasound and: Unequivocal MIBG uptake in tumor Elevated catecholamines in serum or urine No primitive neuroectodermal tumor or primary intracerebral neuroblastoma Such patients referred to protocol GER-HIT90

PATIENT CHARACTERISTICS: Age: Under 21 Other: No serious cerebral trouble No severe concomitant disease, e.g.: No severe congenital malformation No severe organ function abnormality

PRIOR CONCURRENT THERAPY: No prior cytostatic therapy (e.g., for Wilms' tumor) No concurrent therapy

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 1990-07; Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Berthold, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- University of Cologne, Frechen, Germany

REFERENCES:
- [Background] Krams M, Hero B, Berthold F, Parwaresch R, Harms D, Rudolph P. Proliferation marker KI-S5 discriminates between favorable and adverse prognosis in advanced stages of neuroblastoma with and without MYCN amplification. Cancer. 2002 Feb 1;94(3):854-61. PMID 11857322
- [Background] Simon T, Hero B, Dupuis W, Selle B, Berthold F. The incidence of hearing impairment after successful treatment of neuroblastoma. Klin Padiatr. 2002 Jul-Aug;214(4):149-52. doi: 10.1055/s-2002-33179. PMID 12165893
- [Background] Berthold F, Hero B, Kremens B, Handgretinger R, Henze G, Schilling FH, Schrappe M, Simon T, Spix C. Long-term results and risk profiles of patients in five consecutive trials (1979-1997) with stage 4 neuroblastoma over 1 year of age. Cancer Lett. 2003 Jul 18;197(1-2):11-7. doi: 10.1016/s0304-3835(03)00076-4. PMID 12880954
- [Background] von Schweinitz D, Hero B, Berthold F. The impact of surgical radicality on outcome in childhood neuroblastoma. Eur J Pediatr Surg. 2002 Dec;12(6):402-9. doi: 10.1055/s-2002-36952. PMID 12548494
- [Result] Simon T, Hero B, Hunneman DH, Berthold F. Tumour markers are poor predictors for relapse or progression in neuroblastoma. Eur J Cancer. 2003 Sep;39(13):1899-903. doi: 10.1016/s0959-8049(03)00376-9. PMID 12932669
- [Result] Haberle B, Hero B, Berthold F, von Schweinitz D. Characteristics and outcome of thoracic neuroblastoma. Eur J Pediatr Surg. 2002 Jun;12(3):145-50. doi: 10.1055/s-2002-32721. PMID 12101494
- [Result] Hero B, Hunneman DH, Gahr M, Berthold F. Evaluation of catecholamine metabolites, mIBG scan, and bone marrow cytology as response markers in stage 4 neuroblastoma. Med Pediatr Oncol. 2001 Jan;36(1):220-3. doi: 10.1002/1096-911X(20010101)36:13.0.CO;2-6. PMID 11464889